CLINICAL TRIAL: NCT05630495
Title: Validation of an Innovative Neonatal Jaundice Detection System (Picterus) in Indonesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Picterus AS (Industry)
Collaborators: Universitas Airlangga (Other); RSIA Kendangsaru MERR Surabaya (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2018/1608Indonesia2022
Record Dates: First submitted 2022-11-08; First posted 2022-11-29 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-03

CONDITIONS: Jaundice, Neonatal
MeSH Terms: conditions — Jaundice, Neonatal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Enable high qualitative estimation of bilirubin levels in the blood of new-borns (Experimental): In this study we aim to collect data of newborns with wider range of bilirubin levels and additionally measurements of skin color reflectance with a spectrophotometer, to adjust the Picterus JP algorithm and optimize the app performance. This will enable a high qualitative estimation of bilirubin levels in the blood of new-borns of South-East Asian ethnicity and skin type.
  Interventions: Device: Picterus Jaundice Pro

INTERVENTIONS:
Device: Picterus Jaundice Pro — Use Picterus Jaundice Pro, a smartphone app that is used to take photo of the newborns skin, where the Picterus calibration card is place.
  Other Names: Picterus JP

SUMMARY:
The long-term goal of this project is to establish Picterus as a permanent tool to detect NNJ in the healthcare services of Indonesia. Offering early detection and therefore, timely treatment to NNJ, will substantially improve neonatal health and directly work towards the Sustainable Development Goal 3.2.2, reduce neonatal mortality. The study as the following specific subgoals:

* Demonstrate that Picterus system performs accurately in Indonesian newborns
* Ensure that Picterus is in line with users' needs in Indonesia

DETAILED DESCRIPTION:
The long-term goal of this project is to establish Picterus as a permanent tool to detect NNJ in the healthcare services of Indonesia. Offering early detection and therefore, timely treatment to NNJ, will substantially improve neonatal health and directly work towards the Sustainable Development Goal 3.2.2, reduce neonatal mortality. The study as the following specific subgoals:

* Demonstrate that Picterus system performs accurately in Indonesian newborns
* Ensure that Picterus is in line with users' needs in Indonesia

ELIGIBILITY:
Inclusion Criteria:

- Infants born with gestational age ≥37 weeks Birth weight ≥2000g and ≤4500g Age 1 - 14 days

Exclusion Criteria:

- Infants transferred to the pediatric ward for advanced treatment. Infants with a skin rash or other disease that affects the skin where measurements are performed.

Infants that receive or have received phototherapy in the last 24 hours. Infants with an inborn disease

Ages: 1 Day to 14 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2022-12-12 (Actual); Primary Completion 2023-12-15 (Estimated); Study Completion 2024-05-15 (Estimated)

PRIMARY OUTCOMES:
Enable high qualitative estimation of bilirubin levels in the blood of Indonesian newborns | 6 months
  Enable high qualitative estimation of bilirubin levels in the blood of Indonesian newborns using Picterus JP.

SECONDARY OUTCOMES:
Correlation with TcB | 5-10 minutes
  Correlate the estimates of bilirubin levels obtained by Picterus with TcB
Correlation with Tsb and TcB | 1-2 hours
  Correlate the estimates of bilirubin levels obtained by Picterus with TSB and TcB
Picterus JP accuracy in Indonesian newborn | 6 months
  Determine the accuracy of Picterus in Indonesian newborns

CONTACTS AND LOCATIONS:
Overall Officials: Anders Aune, MD,MPH, Study Director — Picterus AS
Locations (2):
- Indonesia (2):
  - Universitas Airlangga Teaching Hospital, Surabaya
  - RSIA Kendangsari MERR hospital, Surabaya

IPD SHARING:
Plan to Share IPD: No